CLINICAL TRIAL: NCT02531919
Title: Chronic Oral Bicarbonate Feasibility Study
Brief Title: Extended Use of Sodium Bicarbonate in Patients With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1300000483
Record Dates: First submitted 2015-08-20; First posted 2015-08-25 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Malignant Neoplasm
Keywords: tumor acidity
MeSH Terms: conditions — Neoplasms | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sodium Bicarbonate (Experimental): Dose concentration of 0.5 g/kg/day
  Interventions: Drug: Sodium Bicarbonate

INTERVENTIONS:
Drug: Sodium Bicarbonate — Given PO
  Other Names: Baking Soda; Bicarbonate of Soda; NaHCO3; Sodium Hydrogen Carbonate

SUMMARY:
This pilot phase I trial studies the safety of long-term use of sodium bicarbonate in patients with cancer. Sodium bicarbonate may neutralize tumor acidity and as a result may inhibit the spread of the tumor to other parts of the body (metastases) and improve survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if the dose concentration of 0.5 g/kg/day sodium bicarbonate is feasible and well tolerated as measured by the proportion of subjects with first evidence of adherence failure.

SECONDARY OBJECTIVES:

I. Determine if the dose concentration of 0.5 g/kg/day sodium bicarbonate is safe for long term consumption (90 days) as measured by blood pressure, resting pulse rate, and basic metabolic panels to assess metabolic alkalosis.

OUTLINE:

PHASE I (RUN-IN/ADJUSTMENT): Patients receive sodium bicarbonate orally (PO) dissolved in water thrice daily (TID) or twice daily (BID) on days 1-10. The dose may be adjusted as necessary.

PHASE II (LONG TERM): Patients continue to receive sodium bicarbonate PO TID or BID for a total of 90 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Any cancer patient enrolled in the study must have a written approval from their oncologist that a notation will be made in the patient's chart for their study participation
* Subject without known cognitive impairment, central nervous system (CNS) metastasis, overt psychosis, major depression, or delirium as noted in the oncology medical record
* Subject with a Karnofsky performance status scale of 80% or greater at time of consent
* Subject has completed initial adjuvant therapy and is not currently receiving or waiting to receive chemotherapy during the next 120 days
* Breast cancer subjects may be enrolled if they are receiving hormonal blockade therapy
* Subject is not enrolled in any other clinical trials
* Subject has a valid working phone number to be contacted with during the study
* Subject must be willing to provide urine specimen for pH measurements during scheduled clinical visits
* Subject must be willing to provide a 3 mL blood sample for metabolic panels during scheduled clinical visits
* Subject does not have uncontrolled hypertension (systolic pressure > 140, diastolic pressure > 90) despite maximal anti-hypertensive therapy
* Subject has healthy renal function: creatinine clearance: 88-128 mL/min; glomerular filtration rate (GFR): > 90 mL/min/1.7m^2 based on standard care results no older than 2 weeks; if no data exist, the subject will need to consent to a blood draw for a basic metabolic panel (which measures creatinine) for verification
* Subject must be informed of the investigational nature of this study and must sign and written informed consent in accordance with institutional and federal guidelines
* Subject is not pregnant or breastfeeding at time of consent; a pregnancy test will be conducted from urine sample on day of consent in premenopausal women
* Subject agrees to use medically approved contraception (ie. condoms, oral contraceptive) if premenopausal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Adherence measured by the time to evidence of adherence failure | 120 days

SECONDARY OUTCOMES:
Assessment of Metabolic Alkalosis by measurement of blood pH from basic metabolic panels | 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Ian Robey, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Medical Center-University Campus, Tucson, Arizona, United States